CLINICAL TRIAL: NCT06897982
Title: One-arm Feasibility and Acceptability Pilot Study of a Community-informed Nutrition Intervention to Recruit, Engage, and Retain Patients Who Are Eligible to Participate in the Diabetes Prevention Program at Two Community Health Centers in Los Angeles
Brief Title: Feasibility of a Nutrition Intervention for Patients With Prediabetes at a Federally Qualified Health Center
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yelba Castellon-Lopez, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004061; 7K23DK129828-03 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prediabetic State; PreDiabetes; Health Knowledge, Attitudes, Practice; Nutrition, Healthy; Acceptability of Health Care; Obesity Prevention
MeSH Terms: conditions — Prediabetic State; Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DPP Clinic Participants (Experimental): A single arm approach with two groups of ten collected a two different time points in the year of the clinic's DPP. These will not be compared to each other they will be used to collect feasibility outcomes data to inform a future pilot randomized study
  Interventions: Behavioral: One-arm feasibility pilot of a nutrition intervention to recruit, engage, and retain DPP participants in the safety-net setting in Los Angeles

INTERVENTIONS:
Behavioral: One-arm feasibility pilot of a nutrition intervention to recruit, engage, and retain DPP participants in the safety-net setting in Los Angeles — This clinical trial incorporates a behavioral intervention as the primary outcome of Aim 3 is to assess the feasibility and acceptability of adding an educational intervention using nutritional demonstrations aligned with the Diabetes Prevention Program (DPP) curriculum among patients who are at-risk for prediabetes. The purpose of this study is to assess if having a nutritional demonstration as part of the DPP would be accepted by clinic DPP patients and hear their perspectives about if this would help them in achieving DPP goals of achieving at least 5% weight loss and implementing sustainable lifestyle changes with healthy eating to reduce their risk of prediabetes. The intervention is designed to encourage healthier eating habits and encourage clinic DPP patients to incorporate this into their daily lives. This study will also determine if it is feasible to incorporate nutritional demonstrations to enhance the existing DPP curriculum

SUMMARY:
The purpose of the study is to assess the feasibility and acceptability of incorporating hands-on nutritional demonstrations to enhance the Diabetes Prevention Program (DPP) curriculum among patients who are at-risk for prediabetes

DETAILED DESCRIPTION:
The purpose of Aim 3 is to assess the feasibility and acceptability of incorporating hands-on nutritional demonstrations to enhance the Diabetes Prevention Program (DPP) curriculum among patients who are at-risk for prediabetes. We will conduct a single arm feasibility study to collect information that will help inform a future pragmatic and fully powered RCT comparing DPP + nutritional intervention and DPP alone. Participants will be recruited from federally qualified health center community clinics with an active DPP course in session. We hypothesize that participants who undergo a 7-week nutritional intervention will not only aid DPP participation and retention but provide participants with the opportunity to apply the nutrition concepts they are actively learning in the DPP in a real-world scenario so that they can incorporate it into their daily lives. Thus, aiding in the DPP's goals of achieving at least 5% weight loss and implementing sustainable lifestyle changes with healthy eating.

A total of 20 participants will be recruited from our partner federally qualified health center, safety-net community clinic sites with an existing DPP: Northeast Valley Health Corporation and AltaMed. We will recruit 2 cohorts of 10 participants each. Participants will be asked to participate in a total 7-week educational intervention using nutritional demonstrations aligned with the DPP curriculum among patients who are at-risk for prediabetes. Healthy cooking demonstrations will be led by a trained community health worker (CHW) with experience teaching about nutrition. The sessions will be co-designed by a registered dietician. Classes will be held at a community resource center with space for conducting cooking demonstrations. Classes will be held in conjunction with the existing DPP curriculum and will be offered as an opportunity to apply what is learned in the DPP curriculum. The cooking demonstrations will be in-person with a virtual option available for participants to join in if they are unable to make it to the class. This aligns with current DPP practices as participants have the option to join DPP classes in combination modality (in-person and via Zoom). The cooking demonstrations will be interactive and designed to provide individuals with prediabetes or who are at high risk of prediabetes, the skills they need to independently prepare healthy, balanced meals that support blood sugar management. The trained CHW and study team will be available to address participant questions or concerns during the 7-week cooking demonstration period. The study team will also conduct weekly check-ins with the participants during this period to collect surveys to measure satisfaction, nutritional knowledge, consumption of fruits and vegetables, and healthy eating habits. Dr. Castellon-Lopez and the study team will use standard surveys and open-ended questions to ensure that we capture the full range of perspectives from all the participants weekly and at the end of the 7-week intervention period, we will conduct audio-recorded interviews with the study participants. As this study does not involve randomization or comparison of different groups receiving different interventions, special methods for randomization are not required. Instead, the study will focus on qualitative and descriptive measures of feasibility and acceptability, such as participant feedback and engagement with nutritional intervention. The sample size was chosen based on the goal of gathering initial data on the intervention's feasibility rather than statistical comparisons or outcome changes. Data analysis will focus on understanding the intervention's feasibility within the existing DPP class structure and the acceptability of the intervention to the participants. As this is a feasibility study, our goal is to collect outcomes to plan for a future fully powered RCT and we do not anticipate having enough power to detect change in outcomes in the current study

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* BMI of 25 or higher (23 or higher if Asian)
* Meet specific blood sugar test criteria indicating prediabetes, such as a fasting plasma glucose level between 110-125 mg/dL or an A1C level between 5.7-6.4%
* Not be diagnosed with type 1 or type 2 diabetes
* Moderate to high risk of having prediabetes or a known diagnosis of prediabetes by their medical provider in the last 12 months.
* Eligible or enrolled in the Diabetes Prevention Program

Exclusion Criteria:

* Younger than 18 years of age
* BMI of less than 25 or higher (or under 23 if Asian)
* Does not meet specific blood sugar test criteria indicating prediabetes, such as a fasting plasma glucose level between 110-125 mg/dL or an A1C level between 5.7-6.4%
* Currently diagnosed with type 1 or type 2 diabetes
* Has not been diagnosed as moderate to high risk of having prediabetes or having a known diagnosis of prediabetes by their medical provider in the last 12 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Retention | Post-Intervention (12-months as DPP is a year-long program)
  The primary outcome of this feasibility study will be retention in the DPP. Retention will be defined as participation in 9 of the 16 core DPP sessions during months 1 through 6 of the DPP. This measure will assess participant completion of the DPP. % retention will be measured at the end of the DPP.

SECONDARY OUTCOMES:
Recruitment Rate of Participants for Nutrition Intervention | Baseline and During Intervention (Weeks 1-7)
  Secondary outcomes of this feasibility study will be to assess the number of DPP patients recruited for this nutrition intervention study. This will be assessed initially at Baseline by total number enrolled and during the intervention (Weeks 1-7) by collecting participant attendance at each weekly nutrition intervention session to see if there is any change in attendance.
Change in Participant Acceptability of the Nutrition Intervention | During & Post-Intervention (Weeks 1-7)
  Secondary outcomes of this feasibility study will be to assess participant acceptability of the nutrition intervention, as defined by satisfaction with the nutrition intervention's cooking demonstration activities. This will be measured via a weekly Likert scale, intervention satisfaction survey. At the end of the intervention (Week 7) participants will participate in a focus group to assess satisfaction and overall acceptability of the nutrition intervention

OTHER OUTCOMES:
Healthy Food Environment Assessment | Pre-Intervention at Baseline in Week 1
  Using the 3-Item Healthy Food Environments Protocol, a self-reported food environment assessment, the study will measure the quality and availability of fresh fruit and vegetables and low-fat products in the local neighborhood. Higher mean scores indicate greater availability of healthy foods in the neighborhood (i.e., low-fat products, fruits, and vegetables).
Change in Food Insecurity | Pre- and Post-intervention (Baseline in Week 1, and Week 7)
  Other outcomes of this feasibility study will collect data on participant experience with food insecurity. This will be evaluated using a 6-Item food Insecurity measure from U.S. Department of Agriculture Economic Research Service.
Change in Self-Efficacy | Pre, During and Post-Intervention (Baseline in Week 1, Week 4, Final session in 7th week)
  Other outcomes of this feasibility study will collect a self-report measure of self-efficacy using a 4-item Brief Self-Efficacy Scale for Healthful Eating
Change in Biometric Data | Pre, During and Post-intervention (Baseline in Week 1, Weekly during 7-wk intervention, Final session in 7th week and at 12 months for DPP end)
  Other outcomes of this feasibility study will collect data on participant weight (this is already collected at DPP classes) HR, sleep hours. The purpose of collecting this data is to assess potential outcomes that should be collected in a future pragmatic and fully powered RCT comparing DPP + nutritional intervention and DPP alone.
Change in Food Consumption Frequency | Pre-Intervention at Baseline, During, and Post-Intervention (Week 1, Week 4 and Week 7)
  Using a self-reported food frequency questionnaire, the study will measure the frequency of specific food and beverage consumption. Participants report how often they consume specific food and beverages using an ordinal response scale ranging from one time per month or less to six or more times per day. Higher scores indicate more frequent consumption.
Change in Dietary Habits | Pre-Intervention and Post-Intervention (Week 1 at Baseline and Week 7)
  The Dietary Screener Questionnaire (DSQ) is a 30-item questionnaire from the National Health and Nutrition Examination Survey (NHANES) 2009-2010 series. The interview includes items about frequency of intake of various food items (per month, daily, etc.).
Change in Quality of Life Indicators | Pre, During and Post-Intervention (Baseline in Week 1, Weekly during 7-wk intervention, Final session in 7th week) and at 12mo
  Other outcomes of this feasibility study will collect a self-reported outcome measure assessing the impact of health on an individual's everyday life to assess quality of life through domains of 1) imitations in physical activities because of health problems 2) Limitations in social activities because of physical or emotional problems 3) Limitations in usual role activities because of physical health problems 4) Bodily pain 5) General mental health (psychological distress and well-being) 6) Limitations in usual role activities because of emotional problems 7) Vitality (energy and fatigue) 8)General health perceptions
Health Literacy | Pre-Intervention at Baseline in Week 1
  Using the Health Literacy Screening Tool - Confidence with Forms, the study will measure participant health literacy at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yelba Castellon-Lopez, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States